CLINICAL TRIAL: NCT03437096
Title: Association Between Postoperative Pain and Venipuncture Pain in Sleeve Gastrectomy Patients
Brief Title: Postoperative Pain and Venipuncture Pain
Acronym: venipuncture
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tokat Gaziosmanpasa University (Other)
Responsible Party: Principal Investigator, fatih altıparmak, Anesthesiology and reanimation, Tokat Gaziosmanpasa University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-KAEK-178
Record Dates: First submitted 2018-02-03; First posted 2018-02-19 (Actual); Last update posted 2018-04-04 (Actual); Status verified 2018-04

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- venipuncture pain (Other): pain during venipuncture
  Interventions: Other: venipuncture pain

INTERVENTIONS:
Other: venipuncture pain — postoperative sleeve gastrectomy patients pain

SUMMARY:
Association between venipuncture pain and postoperative pain

DETAILED DESCRIPTION:
Association will be find between venipuncture pain and postoperative pain in sleeve gastrectomy patients. Also we can study with pain catastrophising scale.

ELIGIBILITY:
Inclusion Criteria:

* sleeve gastrectomy

Exclusion Criteria:

* psychotic illness

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1 (Estimated)
Dates: Start 2018-01-15 (Actual); Primary Completion 2018-05-15 (Estimated); Study Completion 2018-05-16 (Estimated)

PRIMARY OUTCOMES:
numeric rating scale | 3 months
  pain intensity 0 to 10 during venipuncture

CONTACTS AND LOCATIONS:
Overall Officials: Mustafa Süren, Principal Investigator — Gaziosmanpasa University
Locations (1):
- Gaziosmanpasa University, Tokat Province, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided